CLINICAL TRIAL: NCT07182526
Title: Impact of Adding Quercetin or Alpha Lipoic Acid as an Adjuvant Therapy on Clinical and Biochemical Outcomes in a Sample of Iraqi PCOS Patients
Brief Title: Effects of Adding Quercetin or Alpha Lipoic Acid to Usual Care on Symptoms and Blood Markers in Iraqi Women With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Mohammed Mahmood Mohammed, professor, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mustansiriyah University/ 85
Record Dates: First submitted 2025-05-29; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Quercetin; Capsules; Thioctic Acid; Tablets; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quercetin group (Experimental): patients assigned to be treated with metformin 500 mg plus a daily dose of Quercetin 500 mg capsule after meal for three months period.
  Interventions: Drug: Quercetin; Drug: MetFORMIN 500 Mg Oral Tablet
- Alpha lipoic acid group (Experimental): patients assigned to be treated with metformin 500 mg plus a daily dose of Alpha lipoic acid 600mg SR capsule after meal for three months period.
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Tablet; Drug: MetFORMIN 500 Mg Oral Tablet
- Control group (Active Comparator): patients assigned to be treated with metformin 500 mg daily
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet

INTERVENTIONS:
Drug: Quercetin — Quercetin 500 mg capsule daily after meal for three months
  Other Names: Quercetin 500 mg capsule, NOW pharmacetics
  Arms: Quercetin group
Drug: Alpha Lipoic Acid 600 MG Oral Tablet — Alpha lipoic acid 600mg SR capsule daily after meal for three months period.
  Other Names: Alpha lipoic acid 600 mg oral Tablet, Nutricost pharmacetics
  Arms: Alpha lipoic acid group
Drug: MetFORMIN 500 Mg Oral Tablet — metformin 500 mg daily for three months
  Other Names: Glucophage 500 Mg Oral Tablet, Merck pharmacetics

SUMMARY:
This study will investigate whether the addition of Quercetin or Alpha-Lipoic Acid (ALA) to standard metformin therapy can improve symptoms, hormone levels, metabolic health, and quality of life in women with polycystic ovary syndrome (PCOS). Over 3 months, participants will be randomly assigned to one of three groups: metformin alone, metformin plus Quercetin, or metformin plus ALA. Researchers will measure changes in hormones, blood sugar, cholesterol, and antioxidant markers, as well as quality of life and medication adherence. Physical measurements and side effects will also be recorded to assess safety and overall benefit.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if adding Quercetin or Alpha-Lipoic Acid (ALA) to metformin can better treat PCOS symptoms and improve safety, metabolic health, and quality of life in women.

The main questions it aims to answer are:

* Does metformin + Quercetin or metformin + ALA improve hormonal balance (e.g., LH, FSH, testosterone) more than metformin alone?
* Do these combinations enhance glycemic control (fasting glucose, insulin, HOMA-IR), lipid profiles, and oxidative-stress markers (fibulin-1, kisspeptin, SOD1, GPx)?
* How do these regimens affect patient-reported outcomes like quality of life (PCOSQ) and medication adherence?

Researchers will compare three groups to see which regimen yields the greatest improvements:

* Metformin 500 mg daily alone
* Metformin 500 mg + Quercetin 500 mg daily
* Metformin 500 mg + ALA 600 mg SR daily

Participants will:

* Take their assigned oral treatments once daily after a meal for 3 months
* Provide fasting blood samples at baseline and month 3 for hormone, glucose/insulin, lipid, and antioxidant assays
* Complete the PCOSQ quality-of-life questionnaire and the 4-item Morisky adherence scale at both visits
* Undergo physical measurements (weight, BMI, waist/hip circumference, blood pressure) and report any side effects

ELIGIBILITY:
Inclusion Criteria:

* • Newly diagnosed patients should be at reproductive aged from 18-40 years.

  * Patients diagnosed with presence of micro polycystic ovaries at ultrasound.
  * Oligomenorrhea with inter-menstrual intervals longer than 35 days.
  * Clinical or biochemical signs of hyperandrogenism (acne, hirsutism).
  * Normal PRL levels.

Exclusion Criteria:

* • Presence of enzymatic adrenal deficiency and/or other endocrine disease, including diabetes.

  * Other comorbidities (such as hypertension, cardiovascular disease, or hormonal dysfunction).
  * Women who used oral contraceptives, hormonal therapy, or anti-lipidemic drugs.
  * Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hormonal Profile (LH, FSH, Testosterone) from Baseline | Baseline and 3 months after starting assigned treatment
  Serum luteinizing hormone (LH), follicle-stimulating hormone (FSH), and total testosterone levels will be measured in fasting blood samples. Changes from baseline to 3 months will be compared between groups to assess improvement in hormonal balance in women with PCOS.
Change in Glycemic Control Markers (Fasting Glucose, Insulin, HOMA-IR) from Baseline | Baseline and 3 months after starting assigned treatment
  Fasting plasma glucose and insulin will be measured, and the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated. Changes from baseline to 3 months will be compared between groups to evaluate improvements in glycemic control.

SECONDARY OUTCOMES:
Change in Lipid Profile (Total Cholesterol, LDL-C, HDL-C, Triglycerides) from Baseline | Baseline and 3 months after starting assigned treatment
  Fasting lipid panel will be assessed, including total cholesterol, low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglycerides. Changes from baseline to 3 months will be compared between groups.
Change in Oxidative Stress and Related Biomarkers (Fibulin-1, Kisspeptin, SOD1, GPx) from Baseline | Baseline and 3 months after starting assigned treatment
  Serum levels of fibulin-1, kisspeptin, superoxide dismutase 1 (SOD1), and glutathione peroxidase (GPx) will be measured in fasting blood samples. Changes from baseline to 3 months will be compared between groups to assess antioxidant and oxidative stress status.
Change in Quality of Life (PCOSQ Total Score) from Baseline | Baseline and 3 months after starting assigned treatment
  The Polycystic Ovary Syndrome Health-Related Quality of Life Questionnaire (PCOSQ) will be administered. Changes in total score from baseline to 3 months will be compared between groups to evaluate patient-reported well-being.
Change in Medication Adherence (4-Item Morisky Scale Score) from Baseline | Baseline and 3 months after starting assigned treatment
  The 4-item Morisky Medication Adherence Scale will be used to assess adherence to assigned treatment. Changes in score from baseline to 3 months will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Mustansiriyah University/ College of Pharmacy, Baghdad, Karkh, Iraq

IPD SHARING:
Plan to Share IPD: Undecided